CLINICAL TRIAL: NCT06001086
Title: A Multicenter, Open Phase II Clinical Study to Evaluate the Efficacy and Safety of Disitamb Vedotin Combined With Pyrotinib in Previously Untreated Histologically Proven HER2 Positive Early Breast Cancer
Brief Title: A Phase II Clinical Study of Treatment With Disitamb Vedotin Plus Pyrotinib in HER2-positive Early Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230722RC48
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: HER2-positive; RC48
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamb Vedotin combined with pyrotinib (Experimental): Disitamb Vedotin: 2 mg/kg，ivgtt，d1,14/28day/cycle pyrotinib:320mg, oral, every day.
  Interventions: Drug: Disitamb Vedotin ,pyrotinib

INTERVENTIONS:
Drug: Disitamb Vedotin ,pyrotinib — Disitamb Vedotin combined with pyrotinib
  Other Names: Regular Visits

SUMMARY:
Evaluate the efficacy and safety of Disitamb Vedotin combined with pyrotinib in HER2 positive early breast cancer

DETAILED DESCRIPTION:
The main goal of this clinical trial is to evaluate the efficacy of Disitamb Vedotin combined with pyrotinib in previously untreated histologically proven HER2 positive early breast cancer and evaluate the PCR DFS,OS and safety of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 75 years old (at the time of signing the informed consent form), regardless of gender.

2. Subject type and disease characteristics. Histologically confirmed HER2 positive EBC subjects:

1. evaluated as HER2 positive in local laboratories according to ASCOCAP guidelines.
2. Single and multifocal tumors (greater than 1 tumor area limited to the same quadrant as the primary tumor) must be sampled from 1 lesion and laboratory confirmed as HER2 positive.
3. Multicenter tumors (multiple tumors involving more than one breast quadrant) must sample one lesion from each affected quadrant and be confirmed as HER2 positive by the central laboratory.
4. According to ASCOCAP guidelines, tumors are either HR positive or HR negative (ER and PgR negative).
5. Clinical staging at visit (based on breast X-ray or breast MRI evaluation): Stage II-IIIC determined by the AJCC staging system, 8th edition. (f) Lymph node involvement is determined by fine needle aspiration or coarse needle aspiration biopsy (if applicable).

   3. When randomized, ECOG physical fitness status is 0 or 1 point.

   Exclusion Criteria:
   1. Previous history of invasive breast cancer.
   2. Stage IV breast cancer according to AJCC staging system version 8.
   3. Within 3 years, there is any primary malignant tumor, except for fully resected non-melanoma skin cancer or cured in situ disease.
   4. DCIS medical history, except for the subjects who only received Mastectomy
   5. According to the judgment of the researchers, there is evidence of any diseases (such as severe or uncontrolled systemic diseases, including persistent or active infections, uncontrolled hypertension, kidney transplantation and active bleeding diseases, and severe chronic gastrointestinal diseases related to diarrhea) that the researchers consider to be unfavorable for the participants to participate in the study or may affect adherence to the protocol.
   6. Uncontrolled infection requiring intravenous administration of antibiotics, Antiviral drug or antifungal drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response（pCR） | 1 year
  The pCR rate is defined as the proportion of subjects who, after completion of neoadjuvant therapy, showed no evidence of residual invasive lesions in H&E staining in completely excised breast specimens and all sampled local lymph nodes (ypT0/TisypN0) through central evaluation

SECONDARY OUTCOMES:
Disease free survival （DFS) | 3 years
  The time from randomization until disease recurrence or death due to progression of the disease.
Overall Survival（OS） | 5year
  It is defined as the time from the start of treatment to death for any reason.
The Number of Participants Who Experienced Adverse Events (AE) | 1 year
  according to the CTCAE's grading criteria
Patient Report Outcome（PRO） | 3years
  The report is directly obtained from the patient's self-report of their health status, functional status, and treatment experienceThe European O-rganization for Reasearch and Treatment of Cancer（QLQ-C30）、QLQ-BR32，EQ-5D-5L，PRO-CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No